CLINICAL TRIAL: NCT01433276
Title: The Clinical Efficacy and Safety of a Proprietary Solution Containing Hypertonic Sodium Lactate (Totilac®) Infusion for Resuscitation of Patients With Hemorrhagic Shock Due to Multiple Injuries
Brief Title: Efficacy, Safety of Solution Containing Hyperosmolar Sodium Lactate Infusion for Resuscitation of Patients With Hemorrhagic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innogene Kalbiotech Pte. Ltd (Industry)
Responsible Party: Dr Rikrik Ilyas, Director, Innogene Kalbiotech Pte. Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009/IGK-KAL/09
Record Dates: First submitted 2011-08-10; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-08

CONDITIONS: Hemorrhagic Shock
Keywords: Fluid resuscitation; hemorrhagic shock; Totilac; Ringer's; trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Totilac (Experimental)
  Interventions: Drug: Hyperosmolar sodium lactate
- Ringer's lactate (Active Comparator)
  Interventions: Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hyperosmolar sodium lactate — 1st loading : Upto 2 liters of Ringer's lactate, followed by Totilac which was given 5 mL/kgBW/15 minutes, followed by maintenance 2 mL/kgBW/hour for 3 hours
  Other Names: Kalsolac
  Arms: Totilac
Drug: Ringer's lactate — 1st loading : Upto 2 litres of Ringer's lactate, followed by 5 mL/kgBW/15 minutes,followed by maintenance : 2 mL/kgBW/hour for 3 hours
  Other Names: Lactated Ringer's solution
  Arms: Ringer's lactate

SUMMARY:
Indication: Resuscitation in pts with hemorrhagic shock due to multiple injuries

Prospective, open label RCT in pts. with traumatic hemorrhagic shock in RS Hasan Sadikin Hospital, Indonesia.

PI: Dr. Kiki Lukman, PsBD(K), Surgery, RSHS. Co-PI: (late)Prof. Xavier Leverve MD, PhD, Directeur, INSERM-E0221-Bioenergetique Fondamentale et Appliquée Université Joseph Fourier, France

Hemorrhagic shock is a cause of death in trauma.Fluid resuscitation to ensure stable hemodynamics and microcirculation by rapidly restoring circulating plasma volume could be a cornerstone of managing trauma patients. Excessive fluid accumulation particularly in the interstitial tissue should be avoided. Hypertonic solution shows promise in restoring intravascular volume expansion and microcirculation with less fluid infusion in hypovolemic patients. This study investigated efficacy and safety of hyperosmolar Na lactate(Totilac®) for resuscitating traumatic hemorrhagic shock patients.

Patients with multiple injuries with grade III hemorrhagic shock and RTS ≥4 received std initial fluid resuscitation of upto 2 liters of isotonic crystalloid. They also got similar dose of either hyperosmolar Na lactate or ringer's lactate. Hemodynamic status, fluid balance and and safety was recorded during the study.

DETAILED DESCRIPTION:
Trauma is still an important cause of death and disability worldwide.Trauma patients often experience fluid deficits. In addition to apparent blood loss, fluid deficit might also occur secondary to generalized alterations of the endothelial barrier, resulting in diffuse capillary leakage and fluid shift from the intravascular to the interstitial compartment. Severe volume deficits after trauma result in hemorrhagic shock that further leads to the decrease of tissue perfusion, especially to vital organs and inadequate delivery of oxygen and nutrients necessary for normal tissue and cellular function. Subsequently, inadequate and inappropriate management of hemorrhagic shock frequently results in the development of post trauma multiple organ failure which increases the morbidity and mortality of the patients. Consequences of hypovolemic shock (hemorrhagic shock) due to bleeding are one of the major causes of death in trauma patients. Therefore, fluid replacement to reverse shock and to restore perfusion to vital organs appears to be fundamental in the management of the trauma patient, after ensuring an adequate airway, oxygenation and ventilation.

Effective control of hemorrhage and adequate intravenous fluid administration to restore intravascular volume and maintain the tissue perfusion is crucial for saving the patient's life and resuscitation can exacerbate cellular injury caused by hemorrhagic shock, if resuscitation is not performed properly. The type of fluid used for resuscitation plays an important role in this injury pattern. However, when, how and which fluids are ideal in regards to fluid resuscitation remains controversial. The concept that early, aggressive large - volume resuscitation by administration of isotonic crystalloids in volumes 2 to 3 times the estimated blood loss has been widely accepted and practiced; it has even became the standard-of-care adopted by the ATLS for the treatment of trauma casualties (ATLS congress). In patients with prolonged hemorrhagic shock frequently associated with interstitial fluid deficits in addition to intravascular blood volume, resuscitation fluids were needed to replace the intravascular volume loss and replenish interstitial deficits. It has been suggested that aggressive fluid resuscitation improved survival with better function of patient's vital organ patient's with less frequent renal failure. However, aggressive fluid resuscitation can lead to fulminant pulmonary failure "Acute Respiratory Distress Syndrome (ARDS)" and appears as an early cause of death after severe hemorrhage. Moreover, it was observed that aggressive fluid resuscitation in uncontrolled hemorrhagic shock to attempt to increase blood pressure to normal resulted in increased bleeding from injured vessels, hemodynamic decompensation, and increased mortality, and led to cellular injury when compared to no fluid resuscitation or hypotensive resuscitation (permissive hypotension). Therefore a novel resuscitation strategy that overcomes those issues in the near future is still required.

Hyperosmolar solutions of various concentrations (1.8%-7.5%) have been investigated as resuscitation solutions in vitro, as well as animal and clinical studies, with promising results. Clinical and experimental studies have demonstrated that small volume of hypertonic saline solution is able to restore hemodynamics in traumatic shock patients. Small volume of hypertonic solutions stabilize arterial pressure and cardiac output, improve microvascular flow (increases renal, mesenteric, total splanchic and coronary blood flow), control intracranial pressure, with no deleterious effects on immune functions. Moreover, in hemorrhagic shock models, Hyperosmolar solution has immunomodulatory effects including attenuation of immune-mediated cellular injury, modulating the post-trauma immune response, decreasing neutrophil excitation, decreasing inflammation, neutrophil-endothelial binding, lung damage, and bowel injury. This hypertonic solution was more effective than isotonic crystalloids in minimizing the inflammatory response (especially neutrophil cyto-toxicity) and in preventing lung and liver reperfusion injury, as well as in improving intestinal blood flow. Improved survival rate in traumatic hemorrhagic shock patients treated with hypertonic solution were reported in several trials. The beneficial effect of hypertonic saline has been shown related to its hypertonicity characteristic.

A proprietary solution containing hyperosmolar sodium lactate (Totilac) is a hyperosmolar solution with a physiological concentration of potassium chloride and calcium chloride. Totilac with small volume administration during volume deficits in post cardiac surgery patients improves cardiac output, oxygen delivery, urine output, attenuates metabolic acidosis and maintains stable hemodynamic better compared to isotonic crystalloid. Administration of small dose of Totilac in patients with dengue shock syndrome also improved hemodynamic status and microcirculation. High lactate content in this solution offered more benefit in shock patients when compared to other hypertonic solutions as lactate has been known to act as energy substrate in mitochondrion containing cells and can be easily metabolized in hypoxia. Hypertonicity related effects of hyperosmolar sodium lactate solution in addition to lactate effect may offer at least similar benefits in hemorrhagic shock patients, though until now there is no clinical study conducted to prove efficacy of Totilac in hemorrhagic shock. This study aimed to evaluate the efficacy and safety of Totilac as resuscitative fluid regimen in traumatic shock hemorrhagic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years
* Patients with grade III hemorrhagic shock (who fulfilled at least 2 of these following criteria: 1.5-2 L blood loss estimation, MAP <65 mmHg, pulse pressure <20 mmHg, heart rate >120 times/min, respiratory rate 30-40 times/min or urinary output 5-15 ml/hour) due to multiple injuries (simultaneously injuries in two or more organs of the body)
* Survival probability is >50%, predicted by Revised Trauma Score ≥ 4 (scale 0-7.8408)
* Given written informed consent

Exclusion Criteria:

* Patients with burns >20% of body surface area
* Patients with Glasgow Coma Score ≤ 13 (moderate and severe head injury)
* Patients with systemic diseases which were already present before having trauma, such as: cancer, chronic renal failure, liver failure, decompensated heart failure, AIDS (CD4<200/uL) or HIV serology positive with HAAR
* Hemorrhagic shock patients with trias sign: coagulopathy, acidosis and hypothermia that needs blood transfusion immediately
* Patients who were pregnant before having trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Urinary output (UOP) | 3 hours

SECONDARY OUTCOMES:
Blood pressure | 3 hours
Mean arterial pressure | 3 hours
Heart rate | 3 hours
Respiration rate | 3 hours
Glasgow coma scale value | 3 hours
Fluid balance | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Lukman, SpBD(K), Principal Investigator — Department of Surgery, Dr. Hasan Sadikin Hospital, Bandung, Indonesia
Locations (1):
- Department of Surgery, Dr. Hasan Sadikin Hospital, Bandung, Indonesia